CLINICAL TRIAL: NCT00849121
Title: A Pilot Randomized Two-Arm Study of a DNA Vaccine Encoding Prostatic Acid Phosphatase (PAP) in Patients With Non-Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Two-Arm Study of a DNA Vaccine Encoding Prostatic Acid Phosphatase (PAP) in Patients With Non-Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO08802; H-2008-0102 (Other: Institutional Review Board); NCI-2011-00859 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Results first posted 2014-09-11 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
Keywords: Vaccine; pTVG-HP; Prostate Cancer; Castrate Resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intradermal vaccinations of a DNA vaccine encoding PAP, with GM-CSF as an adjuvant given every 2 weeks for the first 12 weeks, then every 12 weeks until disease progression.
  Interventions: Biological: pTVG-HP with rhGM-CSF
- 2 (Experimental): Intradermal vaccinations of a DNA vaccine encoding PAP, with GM-CSF as an adjuvant given every 2 weeks for the first 12 weeks, then given every 2-week, 4-week, or 3-month intervals as dictated by cellular immune response measurement.
  Interventions: Biological: pTVG-HP with rhGM-CSF

INTERVENTIONS:
Biological: pTVG-HP with rhGM-CSF — pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. biweekly for 6 total doses, followed by pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. every 3 months until radiographic disease progression
  Other Names: DNA-based vaccine encoding PAP
  Arms: 1
Biological: pTVG-HP with rhGM-CSF — pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. biweekly for a minimum of 6 total doses, and continuing biweekly until evidence of T-cell immune response, and then following a booster schedule as defined by evidence of T-cell immune response.
  Other Names: DNA-based vaccine encoding PAP
  Arms: 2

SUMMARY:
The investigators are trying to find new methods to treat prostate cancer. The approach is to try to enhance patients' own immune response against the cancer. In this study, the investigators will be testing the safety of a vaccine that may be able to help the body fight prostate cancer.

The vaccine, called pTVG-HP, is a piece of DNA genetic material that contains genetic code for a protein that is made by the prostate gland, called prostatic acid phosphatase (PAP). The vaccine will be given together with a substance called an adjuvant. Adjuvants are typically given with vaccines and can improve the effect of the vaccine. The adjuvant that will be used in this study is called granulocyte-macrophage colony-stimulating factor (GM-CSF).

The main purpose of this study is to find out whether the vaccine generates long-lived immune responses, and whether a better schedule of vaccination can be found by doing frequent laboratory testing for immune responses. The investigators also want to see if the vaccine stimulates any immune reaction against cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Prostate Cancer
* Castrate Resistant Disease with rising PSA despite continuous treatment with orchiectomy or a LHRH agonist
* Rising PSA after treatment and withdrawal of anti-androgen
* Serum Testosterone <50ng/mL
* Normal organ function per laboratory tests

Exclusion Criteria:

* No evidence of immunosuppression or on treatment with immunosuppressive agents
* Cannot have discontinued LHRH agonist treatment (if not previously treated by orchiectomy) within 6 months prior to study entry
* Must not be concurrently taking other medications or supplements with known hormonal effects (other than the LHRH agonist noted above).
* Cannot have any evidence for metastatic disease on bone or CT scan
* Unable or unwilling to undergo two leukapheresis procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03-16 (Actual); Primary Completion 2014-02-17 (Actual); Study Completion 2014-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Tonelli TP, Eickhoff JC, Johnson LE, Liu G, McNeel DG. Long-term follow up of patients treated with a DNA vaccine (pTVG-hp) for PSA-recurrent prostate cancer. Hum Vaccin Immunother. 2024 Dec 31;20(1):2395680. doi: 10.1080/21645515.2024.2395680. Epub 2024 Aug 29. PMID 39208856
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between 3/16/2009 and 4/24/2012 and were recruited from the UW Carbone Cancer Center Clinics
Groups:
- 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12: Intradermal vaccinations of a DNA vaccine encoding PAP, with GM-CSF as an adjuvant given every 2 weeks for the first 12 weeks, then every 12 weeks until disease progression.
  pTVG-HP with rhGM-CSF: pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered intradermally (i.d.) biweekly for 6 total doses, followed by pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered intradermally every 3 months until radiographic disease progression
- 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12: Intradermal vaccinations of a DNA vaccine encoding PAP, with GM-CSF as an adjuvant given every 2 weeks for the first 12 weeks, then given every 2-week, 4-week, or 3-month intervals as dictated by cellular immune response measurement.
  pTVG-HP with rhGM-CSF: pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. biweekly for a minimum of 6 total doses, and continuing biweekly until evidence of T-cell immune response, and then following a booster schedule as defined by evidence of T-cell immune response.
Period: Overall Study
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12: Intradermal vaccinations of a DNA vaccine encoding PAP, with GM-CSF as an adjuvant given every 2 weeks for the first 12 weeks, then every 12 weeks until disease progression.
  pTVG-HP with rhGM-CSF: pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. biweekly for 6 total doses, followed by pTVG-HP (100 µg) with rhGM-CSF (200 µg) administered i.d. every 3 months until radiographic disease progression
- Total: Total of all reporting groups
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Customized [Number; unit: participants]
  40-49 years | 1 | 0 | 1
  60-69 years | 1 | 6 | 7
  70-79 years | 1 | 3 | 4
  80-89 years | 5 | 0 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With > = Grade 2 Autoimmune Events or >=Toxicities at Least Possibly Related to pTVG-HP With GM-CSF Study Treatment.
Description: The number and severity of toxicity incidents occurring between the pre-treatment and the final off-study evaluation will be collected and assigned an attribution. The toxicities observed will be summarized in terms of types and severities by the NCI Common Terminology Criteria version 3 for each study arm. The number of subjects experiencing grade 2 or higher autoimmune events or grade 3 or higher toxicities felt to be at least possibly related to pTVG-HP with GM-CSF study treatment will be compared between the two arms.
Time Frame: From the time the patient begins treatment until 30 days after the last treatment with pTVG-HP vaccine, up to a maximum of 2 years
Measure: Number; unit: participants
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Number analyzed (Participants) | 8 | 9
participants | 1 | 0

2. Primary Outcome: Number of Participants Who Experience at Least a 3-fold Higher PAP-specific T-cell Frequency or Proliferation Index at One Year Compared to Baseline.
Description: The number of patients with a T-cell immune response will be determined for each study arm. An immune response will be defined as a PAP-specific T-cell frequency or proliferation index at 1 year that is at least 3-fold higher than the baseline T-cell frequency or proliferation index.
Time Frame: Baseline and 1 year.
Measure: Number; unit: participants
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Number analyzed (Participants) | 8 | 8
participants | 3 | 6

3. Secondary Outcome: The Number of Participants Who Experience at Least a Two-fold Increase in the PSA Doubling Time During the Treatment Period.
Description: The number of subjects who experience at least a two-fold increase in the PSA doubling time will be documented for each study arm. The PSA doubling time will be calculated using all PSA values obtained starting on Treatment Day 0 and continuing to end of treatment period and compared to the PSA doubling time collected at study entry prior to beginning study treatment.
Time Frame: Starting at Treatment Day 0 and continuing every 4-6 weeks until end of treatment period, an average of 2 years
Measure: Number; unit: participants
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Number analyzed (Participants) | 8 | 9
participants | 3 | 4

4. Secondary Outcome: The Number of Participants Who Are Metastasis-free at One Year.
Description: The number of subjects who are metastatic-free at one year after starting study treatment will be tabulated for each arm. CT Scans and Bone Scans will be obtained at one year to determine whether metastatic disease is present.
Time Frame: one year from study entry
Measure: Number; unit: participants
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Number analyzed (Participants) | 8 | 9
participants | 6 | 6

ADVERSE EVENTS:
Arm/Group | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 (N=8) | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12 (N=9)
Pulmonary Emboli (Vascular disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased C-spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Left hip
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: pTVG-HP With rhGM-CSF Every 3 Months Post Week 12 (N=8) | 2: pTVG-HP With rhGM-CSF Variable Dosing Post Week 12 (N=9)
Allergic reaction (Immune system disorders) | 1 (1) | 2 (2)
Hypertension (Cardiac disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2)
Chills (General disorders) | 3 (4) | 0 (0)
Fever without neutropenia (General disorders) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 8 (47) | 8 (89)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2
Hot flashes (Endocrine disorders) | 1 (1) | 1 (1)
Heart burn (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (4) | 1 (1)
Back pain (General disorders) | 1 (1) | 3 (3)
Headache (General disorders) | 2 (2) | 1 (1)
Chest/thorax pain (General disorders) | 3 (5) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pain neck (General disorders) | 2 (2) | 0 (0)
Edema (General disorders) | 2 (2) | 0 (0)
Creatinine (Investigations) | 1 (1) | 1 (1)
Sensory (Nervous system disorders) | 0 (0) | 1 (1) — Cramps to hands and feet
Bradcardia (Cardiac disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 2 (2)
Pain Bone (General disorders) | 2 (6) | 4 (4)
Abdominal bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breast tenderness (General disorders) | 0 (0) | 1 (1)
Vision change (Eye disorders) | 1 (1) | 0 (0) — hazy vision
Pain--other (General disorders) | 1 (1) | 0 (0) — testicle pain
Pain--abdomen (General disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Burning on urination
Urinary--other (Renal and urinary disorders) | 1 (1) | 1 (1) — Slow urine stream/dribbling

LIMITATIONS AND CAVEATS:
Of the 17 participants enrolled, 16 received at least 6 initial immunizations with pTVG-HP vaccine and were deemed evaluable to be assessed for outcome measure 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes